CLINICAL TRIAL: NCT02030080
Title: A Randomized Trial of Behavioral Economic Interventions to Improve Physical Activities: Framing vs Incentives
Brief Title: Way to Be Active IV (Framing vs Incentives)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 819371
Record Dates: First submitted 2013-12-20; First posted 2014-01-08 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Sedentary Lifestyle
Keywords: Pedometers; Walking; Financial incentives; Sedentary lifestyle; Behavioral economics
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Feedback 50th Percentile (Active Comparator): At the end of each week, participants will be told the average daily step count for their team for the previous week. They will also be told the average for the 50th percentile in their arm.
  Interventions: Behavioral: Teams; Behavioral: Daily Feedback
- Feedback 75th Percentile (Experimental): At the end of each week, participants will be told the average daily step count for their team for the previous week. They will also be told the average for the 75th percentile in their arm.
  Interventions: Behavioral: Teams; Behavioral: Framing of feedback; Behavioral: Daily Feedback
- Feedback 50th Percentile + Lottery (Experimental): At the end of each week, participants will be told the average daily step count for their team for the previous week. They will also be told the average for the 50th percentile in their arm. If their team's average daily step count is ≥ 7000 steps, they'll be eligible to collect winnings from a weekly lottery. Teams whose average daily step count is less than 7000 will receive messages about how much they would have won had the team met its goal.
  Interventions: Behavioral: Financial incentives; Behavioral: Teams; Behavioral: Daily Feedback
- Feedback 75th Percentile + Lottery (Experimental): At the end of each week, participants will be told the average daily step count for their team for the previous week. They will also be told the average for the 75th percentile in their arm. If their team's average daily step count is ≥ 7000 steps, they'll be eligible to collect winnings from a weekly lottery. Teams whose average daily step count is less than 7000 will receive messages about how much they would have won had the team met its goal.
  Interventions: Behavioral: Financial incentives; Behavioral: Teams; Behavioral: Framing of feedback; Behavioral: Daily Feedback

INTERVENTIONS:
Behavioral: Financial incentives
  Arms: Feedback 50th Percentile + Lottery; Feedback 75th Percentile + Lottery
Behavioral: Teams
Behavioral: Framing of feedback
  Arms: Feedback 75th Percentile; Feedback 75th Percentile + Lottery
Behavioral: Daily Feedback — Participants will be given daily feedback on whether or not they walked 7000 steps or more the day before.

SUMMARY:
Employers are increasingly looking for opportunities to motivate sedentary employees to become more physically active. Workplace walking programs have had mixed success and typically show most improvement among participants that are already fairly active at a baseline. The goal of this study is to determine whether a financial incentive program can motivate sedentary employees to increase the number of steps they walk per day to meet a minimum threshold.

The primary outcome measure is the proportion of days a minimum activity of 7000 steps or more is achieved. Outcomes will be assessed each week for 3 months using incentives followed by 3 months of follow-up without incentives. Secondary outcomes will include the average steps walked per day.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18.
* Participant will need an iPhone or Android smartphone to be able to use the Moves App for tracking steps

Exclusion Criteria:

* Pregnant or lactating
* Currently participating in another physical activity study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, MBA, Study Director — University of Pennsylvania; Kevin Volpp, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Patel MS, Volpp KG, Rosin R, Bellamy SL, Small DS, Fletcher MA, Osman-Koss R, Brady JL, Haff N, Lee SM, Wesby L, Hoffer K, Shuttleworth D, Taylor DH, Hilbert V, Zhu J, Yang L, Wang X, Asch DA. A Randomized Trial of Social Comparison Feedback and Financial Incentives to Increase Physical Activity. Am J Health Promot. 2016 Jul;30(6):416-24. doi: 10.1177/0890117116658195. Epub 2016 Jul 15. PMID 27422252

RESULTS

PARTICIPANT FLOW:
Groups:
- Feedback 50th Percentile: At the end of each week, participants will be told the average daily step count for their team for the previous week. They will also be told the average for the 50th percentile in their arm.
  Teams
  Daily Feedback: Participants will be given daily feedback on whether or not they walked 7000 steps or more the day before.
- Feedback 75th Percentile: At the end of each week, participants will be told the average daily step count for their team for the previous week. They will also be told the average for the 75th percentile in their arm.
  Teams
  Framing of feedback
  Daily Feedback: Participants will be given daily feedback on whether or not they walked 7000 steps or more the day before.
- Feedback 50th Percentile + Lottery: At the end of each week, participants will be told the average daily step count for their team for the previous week. They will also be told the average for the 50th percentile in their arm. If their team's average daily step count is ≥ 7000 steps, they'll be eligible to collect winnings from a weekly lottery. Teams whose average daily step count is less than 7000 will receive messages about how much they would have won had the team met its goal.
  Financial incentives
  Teams
  Daily Feedback: Participants will be given daily feedback on whether or not they walked 7000 steps or more the day before.
- Feedback 75th Percentile + Lottery: At the end of each week, participants will be told the average daily step count for their team for the previous week. They will also be told the average for the 75th percentile in their arm. If their team's average daily step count is ≥ 7000 steps, they'll be eligible to collect winnings from a weekly lottery. Teams whose average daily step count is less than 7000 will receive messages about how much they would have won had the team met its goal.
  Financial incentives
  Teams
  Framing of feedback
  Daily Feedback: Participants will be given daily feedback on whether or not they walked 7000 steps or more the day before.
Period: Overall Study
Arm/Group | Feedback 50th Percentile | Feedback 75th Percentile | Feedback 50th Percentile + Lottery | Feedback 75th Percentile + Lottery
Started | 100 (25 teams) | 64 (16 teams) | 80 (20 teams) | 44 (11 teams)
Completed | 100 | 64 | 80 | 42
Not Completed | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Feedback 50th Percentile | Feedback 75th Percentile | Feedback 50th Percentile + Lottery | Feedback 75th Percentile + Lottery | Total
Number analyzed (Participants) | 100 | 64 | 80 | 42 | 286
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.9 (12.2) | 43.1 (10.5) | 40.7 (12.2) | 40.8 (13.2) | 41.3 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 48 | 69 | 36 | 229
  Male | 24 | 16 | 11 | 6 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 65 | 49 | 50 | 28 | 192
  African American non-Hispanic | 21 | 11 | 15 | 11 | 58
  Other non-Hispanic | 13 | 1 | 12 | 3 | 29
  Hispanic | 1 | 3 | 3 | 0 | 7
Education [Count of Participants; unit: Participants]
  Less than college | 6 | 6 | 4 | 4 | 20
  Some college | 16 | 22 | 16 | 8 | 62
  College graduate | 78 | 36 | 60 | 30 | 204
Marital status [Count of Participants; unit: Participants]
  Single | 36 | 25 | 30 | 14 | 105
  Married | 55 | 35 | 39 | 24 | 153
  Other | 9 | 4 | 11 | 4 | 28
Annual household income [Count of Participants; unit: Participants]
  Less than $50,000 | 19 | 13 | 13 | 8 | 53
  $50,000-$100,000 | 31 | 17 | 28 | 20 | 96
  Greater than $100,000 | 35 | 30 | 29 | 12 | 106
  Missing Data | 15 | 4 | 10 | 2 | 31
Number of Participants with iPhone smartphone [Count of Participants; unit: Participants] | 71 | 48 | 56 | 34 | 209
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 29 (7.4) | 28.7 (6.1) | 27.5 (5.8) | 28.5 (6.2) | 28.4 (6.5)
Physical activity in the last 7 days (MET-min) [Median (Inter-Quartile Range); unit: Metabolic equivalent minutes (MET-min)] — The International Physical Activity Questionnaire (IPAQ) was used to calculate the number of metabolic equivalent minutes (MET-min) per participant in the most recent 7 days. The MET is a physiologic measure of energy expenditure, with light-intensity activities having an MET <3, moderate-intensity activities having an MET of 3 to 6, and more vigorous-intensity activities with an MET>6.
  Metabolic equivalent minutes (MET-min) | 4698.0 [2424.0 to 7740.0] | 4702.5 [2914.5 to 8071.5] | 4186.0 [1711.5 to 7173.0] | 3630.0 [2208.0 to 9588.0] | 4533.3 [2329.5 to 7929.0]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Days a Participant Walks 7000 Steps or More
Description: The primary outcome measure is the proportion of days a minimum activity of 7000 steps or more is achieved. Outcomes will be assessed each week for 3 months using incentives followed by 3 months of follow-up without incentives. Below we report the highest mean proportions found.
Time Frame: Throughout 6-month study
Measure: Mean (95% Confidence Interval); unit: Mean proportion
Arm/Group | Feedback 50th Percentile | Feedback 75th Percentile | Feedback 50th Percentile + Lottery | Feedback 75th Percentile + Lottery
Number analyzed (Participants) | 100 | 64 | 80 | 42
Mean proportion | 0.30 [0.21 to 0.38] | 0.27 [0.17 to 0.37] | 0.45 [0.35 to 0.54] | 0.38 [0.25 to 0.50]

2. Secondary Outcome: Average Number of Steps Per Day
Description: Secondary outcomes include average number of steps per day during the incentive period (first 3 months) and follow-up period (second 3 months).
Time Frame: Throughout the 6-month study
Measure: Mean (95% Confidence Interval); unit: Mean daily step counts
Arm/Group | Feedback 50th Percentile | Feedback 75th Percentile | Feedback 50th Percentile + Lottery | Feedback 75th Percentile + Lottery
Number analyzed (Participants) | 100 | 64 | 80 | 42
Mean daily step counts | 5146 [4472 to 5820] | 4676 [3833 to 5518] | 6032 [5278 to 6785] | 5432 [4415 to 6448]

ADVERSE EVENTS:
Arm/Group | Feedback 50th Percentile | Feedback 75th Percentile | Feedback 50th Percentile + Lottery | Feedback 75th Percentile + Lottery
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/64 | 0/80 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/64 | 0/80 | 0/42
Other Adverse Events (participants affected / at risk) | 0/100 | 0/64 | 0/80 | 0/42

LIMITATIONS AND CAVEATS:
Participants are from single location and their activity was not tracked when not carrying smartphones. Randomization resulted in uneven # of participants; potentially limiting power for arms with < 70 subjects. Did not have baseline data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No